CLINICAL TRIAL: NCT01516970
Title: HIV Postexposure Prophylaxis With Darunavir/r (PEPDar)
Brief Title: Human Immunodeficiency Virus (HIV) Postexposure Prophylaxis (PEP) With Darunavir/Ritonavir (DRV/r)
Acronym: PEPDar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018349; TMC114IFD3004 (Other: Janssen-Cilag G.m.b.H, Germany); 2011-001303-13 (EudraCT Number)
Record Dates: First submitted 2011-10-11; First posted 2012-01-25 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus (HIV) Post exposure prophylaxis; DRV/r; Occupational injury; Non-occupational exposure; Prezista; Darunavir/r
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Occupational Injuries | interventions — Darunavir; Ritonavir; Lopinavir; lopinavir-ritonavir drug combination; Zidovudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- DRV/r with 2 NRTIs (Experimental): DRV/r 800/100 mg q.d. with 2 NRTIs: darunavir (800 mg) in combination with low-dose ritonavir (100 mg) administered once a day for at least 28 days and a maximum of 30 days along with 2 nucleoside/nucleotide analogue reverse transcriptase inhibitors (NRTIs).
  Interventions: Drug: Darunavir/Ritonavir (DRV/r); Drug: NRTIs
- Comparator standard of care HIV PEP (Active Comparator): Comparator standard of care HIV PEP (as per German-Austrian Guidelines): Administration of the standard of care HIV PEP (postexposure prophylaxis) consisting of 2 NRTIs plus third partner.
  Interventions: Drug: Lopinavir in fixed combination with Ritonavir; Drug: Zidovudine; Drug: NRTIs; Drug: Efavirenz

INTERVENTIONS:
Drug: Darunavir/Ritonavir (DRV/r) — Darunavir (DRV) type=exact number, unit=mg, number=800, form=tablet, route=oral use. Tablet is taken once a day, for 28 days; Ritonavir (r) type=exact number, unit=mg, number=100, form=tablet, route=oral use. Tablet is taken once a day, for at least 28 days and a maximum of 30 days.
  Arms: DRV/r with 2 NRTIs
Drug: Lopinavir in fixed combination with Ritonavir — type=exact number, unit=mg, number=400/100, form=tablet, route=oral use. Tablet is taken once or twice a day, for at least 28 days and a maximum of 30 days.
  Other Names: Kaletra
  Arms: Comparator standard of care HIV PEP
Drug: Zidovudine — type=exact number, unit=mg, number=250, form=tablet, route=oral use. Tablet is taken twice a day, for at least 28 days and a maximum of 30 days.
  Other Names: Retrovir
  Arms: Comparator standard of care HIV PEP
Drug: NRTIs — The NRTIs (including tenofovir/emtricitabine [Truvada], lamivudine/zidovudine [Combivir]) will be administered as per the individual Summary of Product Characteristics (SmPCs) at the discretion of either the treating physician or Investigator.
Drug: Efavirenz — type=exact number, unit=mg, number=600, form=tablet, route=oral use. Tablet is taken once a day, for at least 28 days and a maximum of 30 days.
  Other Names: Sustiva
  Arms: Comparator standard of care HIV PEP

SUMMARY:
The primary purpose of this study is to assess the rate of early discontinuation from randomized Human Immunodeficiency Virus (HIV) Postexposure Prophylaxis (PEP) for any reason other than confirmation of the negative HIV infection status of the index person in patients receiving HIV PEP for at least 28 and a maximum of 30 days.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), open-label (all people involved know the identity of the intervention), active-controlled (patients are assigned to either a recognized effective treatment or the study medication), parallel-group (each treatment group will be treated at the same time), multicenter study comparing DRV/r PEP (DRV/r administered with 2 NRTIs selected at the discretion of the investigator) to standard of care PEP (as per German-Austrian guidelines) in patients at risk of HIV infection due to HIV exposure through occupational injury and non-occupational exposure. This study consists of screening period, treatment period and a follow up period. HIV PEP will be administered for a total of at least 28 days and maximum of 30 days during treatment period, including any prestudy HIV PEP initiated before screening. Approximately 318 patients will be screened and enrolled to ensure that at least 131 patients are randomly assigned to receive DRV/r PEP or standard of care PEP. Safety will be evaluated during the entire study period. Data relating to a patient's functional impairment in conjunction with HIV PEP will be collected on Day 1 as baseline data, and further on Days 14 and 28 as well as at Month 3.

ELIGIBILITY:
Inclusion Criteria:

* Occupational injury and non-occupational exposure with documented human immunodeficiency virus (HIV) exposure, or potential for HIV exposure
* Indication for HIV postexposure prophylaxis (PEP), as determined by the treating physician and/or the investigator
* Women must be: postmenopausal (for at least 2 years), surgically sterile, using oral contraceptives
* Willing to continue HIV PEP for 28 days

Exclusion Criteria:

* Positive HIV rapid test
* History of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastro intestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Pregnant or breast-feeding
* Any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2011-11-25 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (17):
- Germany (17):
  - Berlin
  - Bonn
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Erlangen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Magdeburg
  - Mainz
  - Mannheim
  - München
  - Regensburg
  - Stuttgart
  - Ulm

RESULTS

PARTICIPANT FLOW:
Groups:
- Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP): Darunavir (800 milligram [mg]) in combination with low-dose ritonavir (100 mg) administered once a day for at least 28 days and a maximum of 30 days along with 2 nucleoside/nucleotide analogue reverse transcriptase inhibitors (NRTIs). The NRTIs (including tenofovir/emtricitabine [Truvada] was administered as per the individual Summary of Product Characteristics (SmPCs) at the discretion of either the treating physician or Investigator.
- Standard of Care Postexposure Prophylaxis (SOCPEP): Standard of care human immunodeficiency virus (HIV) PEP (as per German-Austrian Guidelines): Administration of the standard of care HIV PEP (postexposure prophylaxis) consisting of 2 NRTIs plus third partner. Lopinavir in combination with low-dose ritonavir (LPV/r) [Kaletra] was combined with following NRTIs: TDF (tenofovir)/ FTC (emtricitabine) [Truvada], AZT (zidovudine)/3TC (lamivudine) [Combivir]) and ABC (Abacavir)/ 3TC (Lamivudine) administered as per the individual SmPCs at the discretion of either the treating physician or Investigator.
Period: Overall Study
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Started | 159 | 153
Completed | 141 | 132
Not Completed | 18 | 21
Not completed — Lost to Follow-up | 7 | 8
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 9 | 7

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of randomized HIV PEP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP) | Total
Number analyzed (Participants) | 159 | 153 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (9.2) | 32.3 (9.3) | 33.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 131 | 125 | 256

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Discontinuation From Randomized Human Immunodeficiency Virus Postexposure Prophylaxis (HIV PEP)
Description: Number of participants with early discontinuation from randomized HIV PEP for any reason other than confirmation of the negative HIV infection status of the index person in participants receiving HIV PEP for at least 28 days and a maximum of 30 days was assessed. Per protocol (PP) population included all participants in modified intention-to-treat (mITT [defined as all participants who were assigned to receive randomized HIV PEP and were not discontinued due to confirmation of the negative HIV infection status of the index person]) excluding participants with: No indication for HIV PEP; Initiation of PEP >72 hours after injury; Discontinuation of HIV PEP due to confirmation of HIV negative status of index person and if index person bears resistant virus against HIV PEP components prescribed; incorrect HIV PEP; no intake of medication.
Time Frame: Up to 30 days
Population: Analysis was performed on PP population.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Standard of Care Postexposure Prophylaxis (SOCPEP): Standard of care human immunodeficiency virus (HIV) PEP (as per German-Austrian Guidelines): Administration of the standard of care HIV PEP (postexposure prophylaxis) consisting of 2 NRTIs plus third partner. Lopinavir in combination with low-dose ritonavir (LPV/r) [Kaletra] was combined with following NRTIs: TDF (tenofovir)/ FTC (emtricitabine) [Truvada], AZT (zidovudine)/3TC (lamivudine) [Combivir]) and ABC (Abacavir)/ 3TC (Lamivudine) administered as per the individual Summary of Product Characteristics (SmPCs) at the discretion of either the treating physician or Investigator.
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Number analyzed (Participants) | 155 | 150
participants | 10 [3.5 to 11.5] | 15 [6.2 to 15.8]
Statistical Analysis 1: Comparison: Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) vs Standard of Care Postexposure Prophylaxis (SOCPEP); Test type: Superiority or Other; p = 0.2434, Cochran-Mantel-Haenszel — The discontinuation rates were compared with a statistical test (Cochran-Mantel-Haenszel [CMH]-Test) with p-value: 0.2434

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined to be non-treatment-emergent if the onset date of the AE was clearly before the date of first HIV PEP administration, otherwise it is considered treatment-emergent.
Time Frame: Up to Month 3
Population: The safety population included all participants who received at least 1 dose of randomized HIV PEP.
Measure: Number; unit: participants
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Number analyzed (Participants) | 159 | 153
participants | 131 | 125
Statistical Analysis 1: Comparison: Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) vs Standard of Care Postexposure Prophylaxis (SOCPEP); Test type: Superiority or Other; p = 0.8839, Fisher Exact — The percentage of participants with TEAEs were compared with a statistical test (Fisher's Exact Test) with p-value: 0.8839

3. Secondary Outcome: Worst Sheehan Disability Scale (SDS) Score for the Safety Population
Description: The Sheehan Disability Scale (SDS) assesses functional impairment in 3 inter-related domains: work/school, social and family life, using a rating scale for each item ranging from 0 (not at all) to 10 (extremely).
Time Frame: Month 3
Population: The safety population included all participants who received at least 1 dose of randomized HIV PEP.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Number analyzed (Participants) | 159 | 153
units on a scale
  Impairment in work/school/studies | 2.566 (2.775) | 3.503 (2.940)
  Impairment in social life | 2.465 (2.594) | 3.464 (2.786)
  Impairment in family life | 2.226 (2.624) | 2.954 (2.713)

4. Secondary Outcome: Percentage of Participants Who Developed Detectable HIV Antibodies
Description: Seroconversion rate of HIV antibodies while receiving HIV PEP evaluated as the percentage of participants who developed detectable HIV antibodies (defined as positive) and percentage of participants who had not developed detectable HIV antibodies (defined as negative). Per protocol (PP) population included all participants in mITT (defined as all participants who were assigned to receive randomized HIV PEP and were not discontinued due to confirmation of the negative HIV infection status of the index person) excluding participants with: No indication for HIV PEP; Initiation of PEP >72 hours after injury; Discontinuation of HIV PEP due to confirmation of HIV negative status of index person and if index person bears resistant virus against HIV PEP components prescribed; incorrect HIV PEP; no intake of medication.
Time Frame: At Month 3
Population: Analysis was performed on PP population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Number analyzed (Participants) | 138 | 133
percentage of participants
  Negative | 99.3 | 100
  Positive | 0.7 | 0

ADVERSE EVENTS:
Time Frame: Up to Month 3
Description: The safety population included all participants who received at least 1 dose of randomized HIV PEP.
Arm/Group | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) | Standard of Care Postexposure Prophylaxis (SOCPEP)
Serious Adverse Events (participants affected / at risk) | 1/159 | 0/153
Other Adverse Events (participants affected / at risk) | 96/159 | 111/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) (N=159) | Standard of Care Postexposure Prophylaxis (SOCPEP) (N=153)
Depression (Psychiatric disorders) | 1 | 0 — The only serious adverse event observed in the DRV/r arm was a hospitalization due to an unrelated depression.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir/Ritonavir Postexposure Prophylaxis (DRV/r PEP) (N=159) | Standard of Care Postexposure Prophylaxis (SOCPEP) (N=153)
Dizziness (Nervous system disorders) | 6 | 2
Dysgeusia (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 19 | 8
Asthenia (General disorders) | 5 | 1
Fatigue (General disorders) | 21 | 28
Sleep Disorder (Psychiatric disorders) | 0 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 14 | 11
Diarrhoea (Gastrointestinal disorders) | 45 | 76
Flatulence (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 24 | 41
Vomiting (Gastrointestinal disorders) | 10 | 9
Rash (Skin and subcutaneous tissue disorders) | 7 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.